CLINICAL TRIAL: NCT02386995
Title: Comparison of Bispectral Index and Entropy Monitoring in Patients Undergoing Internalization of Deep Brain Simulation
Brief Title: BIS and Entropy in Deep Brain Simulation
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Lashmi Venkatraghavan, Dr., University Health Network, Toronto
Other Study IDs: 13-6060
Record Dates: First submitted 2013-11-28; First posted 2015-03-12 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Movement Disorders; Depth of Anesthesia Monitors
Keywords: depth of anesthesia monitors; deep brain stimulation
MeSH Terms: conditions — Movement Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BIS and Entropy monitoring: Depth of anesthesia monitoring (BIS and entropy) are compared with standard clinical monitoring in patients with deep brain stimulators inserted at internalization whilst they are having a general anesthesia.
  Interventions: Device: BIS monitor; Device: Entropy monitor

INTERVENTIONS:
Device: BIS monitor — Both types of depth of anesthesia monitoring (BIS and entropy- electrodes) are applied on patients together with standard monitoring (heart rate, blood pressure, respiratory rate). The two different types of depth of anesthesia monitoring are then compared.
Device: Entropy monitor — Both types of depth of anesthesia monitoring (BIS and entropy- electrodes) are applied on patients together with standard monitoring (heart rate, blood pressure, respiratory rate). The two different types of depth of anesthesia

SUMMARY:
The main objective of the study is to determine whether depth of anesthesia (DOA) monitoring such as Bispectral Index (BIS) and entropy are accurate in patients with neuro-psychological conditions such as Parkinson's disease by comparing these monitoring with standard clinical monitoring like heart rate, blood pressure and respiratory rate.

DETAILED DESCRIPTION:
Deep brain simulation (DBS) is an increasingly popular treatment for movement and psychiatric disorders such as Parkinson's disease and dystonia. These patients are quite sensitive to anesthetics and use of depth of anesthesia monitors are often needed to titrate the anesthetics. The calibration of BIS and entropy monitors has been done only on subjects with no neurological diseases. The investigators plan to record BIS and entropy readings during general anesthesia (GA) for the internalization of DBS electrodes. This would be useful as there are very few studies in this subset of patients with regards to DOA monitoring. Ashraf argued that the EEG may be altered under these circumstances and hence produce invalid BIS readings. Pemberton et al. studied patients undergoing tumour surgery using a sleep- awake-sleep anaesthesia technique. They found a poor correlation between BIS values and the observer's assessment of anesthesia level, suggesting that BIS is not a reliable tool for patients with brain abnormalities. The purpose of this study was to investigate whether BIS and entropy are helpful in titrating DOA in patients undergoing neurosurgical procedures or suffering from neurological diseases as they were frequently excluded from validation studies of the BIS monitoring device.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients older than 18 years of age scheduled for elective internalisation of DBS electrodes under general anesthesia.

Exclusion Criteria:

* lack of informed consent
* language barrier
* those that are transferred to an intensive care unit postoperatively.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having a general anesthesia post DBS insertion for the internalization of DBS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lashmi Venkatraghavan, Principal Investigator — University Health Network, Toronto Western Hospital; Pirjo Manninen, Principal Investigator — University Heath Network, Toronto Western Hospital; Audrey MY Tan, Principal Investigator — University Heath Network, Toronto Western Hospital
Locations (1):
- University Heath Network, Toronto Western Hospital, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BIS and Entropy Monitoring
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Demographic data values are presented as (mean±SD)
Arm/Group | BIS and Entropy Monitoring
Number analyzed (Participants) | 30
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 58.4 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Bispectral (BIS) and Response Entropy (RE) Indices
Description: The trends of Bispectral (BIS) and Response entropy (RE) at different study time points.
  Bispectral (BIS) and Response entropy (RE) values range from 0 (absence of brain activity) to 100 (fully awake state).
  Values below 40 indicate deep anesthesia, values from 40 to 60 optimal and above 60 but below 90 inadequate anesthesia.
Time Frame: One day
Population: Correlation analysis between BIS and RE from pre-induction time (T1) until the surgical closure time (T9) Bispectral (BIS) and Response entropy (RE) values range from 0 (absence of brain activity) to 100 (fully awake state).
  Values below 40 indicate deep anesthesia, values from 40 to 60 optimal and above 60 but below 90 inadequate anesthesia.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Bispectral Index BIS: The trends of Bispectral index (BIS) at different study time points (T)
- Response Entropy Index: The trends of Response Entropy index (RE) at different study time points (T)
Arm/Group | Bispectral Index BIS | Response Entropy Index
Number analyzed (Participants) | 30 | 30
units on a scale
  T1 Awake (preinduction) | 96 (1) | 96 (3)
  T2 Loss of response to speech | 65 (4) | 77 (9)
  T3 Loss of eyelash reflex | 59 (5) | 63 (6)
  T4 Intubation | 44 (4) | 53 (5)
  T5 Knife to skin | 44 (2) | 44 (5)
  T6 Maintenance (prior to tunneling) | 40 (4) | 33 (4)
  T7 Tunneling in the neck | 36 (6) | 32 (5)
  T8 Start of skin closure | 40 (6) | 37 (6)
  T9 End of skin closure | 42 (8) | 49 (9)
  T10 Anaesthetic agent turned off | 66 (7) | 59 (6)
  T11 Obeying commands | 87 (3) | 89 (6)
  T12 Extubation | 92 (3) | 93 (4)
  T13 Post-extubation | 93 (3) | 96 (2)

ADVERSE EVENTS:
Time Frame: one day
Arm/Group | BIS and Entropy Monitoring
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes